CLINICAL TRIAL: NCT07124273
Title: The Effect of Dental Anxiety on the Success of Mandibular Anesthesia in Mandibular Molar Teeth With Symptomatic Irreversible Pulpitis: A Prospective Clinical Study
Brief Title: Effect of Dental Anxiety on Mandibular Anesthesia Success
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: KutahyaHSU-3
Record Dates: First submitted 2025-08-01; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Dental Anxiety; Symptomatic Irreversible Pulpitis
Keywords: Dental Anxiety; Local Anesthesia Failure; Salivary Cortisol; Symptomatic Irreversible Pulpitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Anxiety Group (Experimental): Participants with Modified Dental Anxiety Scale (MDAS) scores less than 10.
  Interventions: Procedure: Standardized Mandibular Anesthesia Protocol
- Moderate-High Anxiety Group (Experimental): Participants with MDAS scores of 11 or higher, including those with dental phobia (MDAS > 19).
  Interventions: Procedure: Standardized Mandibular Anesthesia Protocol

INTERVENTIONS:
Procedure: Standardized Mandibular Anesthesia Protocol — Participants receive an inferior alveolar nerve block (IANB) using 1.8 ml 4% articaine with 1:100,000 epinephrine (Ultracaine DS Forte) via a 27-gauge dental needle, followed by buccal and lingual infiltration anesthesia after 5 minutes. Topical 10% lidocaine spray is applied prior to injection. All procedures are performed by the same clinician between 09:00-12:00. Salivary cortisol, pulse oximetry, and pain assessments are conducted before and after the anesthesia.

SUMMARY:
The goal of this clinical trial is to evaluate the effect of dental anxiety on the success of mandibular anesthesia in patients with symptomatic irreversible pulpitis in mandibular molar teeth.

The main questions it aims to answer are:

Does dental anxiety influence the success rate of inferior alveolar nerve block (IANB)? Is there a correlation between salivary cortisol levels and anesthesia outcomes in anxious patients?

Researchers will compare two groups of patients based on their Modified Dental Anxiety Scale (MDAS) scores:

Low/No anxiety group (MDAS < 10) Moderate to high anxiety group (MDAS ≥ 11, including those with dental phobia)

Participants will:

Rate their pre-treatment pain using the Heft-Parker Visual Analog Scale (HP-VAS) Provide salivary samples for cortisol measurement before and after anesthesia Undergo standardized mandibular anesthesia protocols (IANB and buccal-lingual infiltration) Report pain during treatment using the HP-VAS Undergo monitoring of SpO₂ and pulse via pulse oximetry To control for cortisol fluctuations and circadian rhythm, all procedures and saliva collections will occur between 09:00-12:00. Participants will be asked to avoid food for at least 2 hours prior, and refrain from caffeine, alcohol, smoking, or heavy exercise for at least 24 hours before treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65 years
* Systemically healthy individuals who agree to participate in the study
* Mandibular molar teeth diagnosed with symptomatic irreversible pulpitis requiring root canal treatment
* Teeth with closed apex and no periapical lesions visible radiographically
* Periodontally healthy teeth according to Glickman's criteria, with probing depth ≤ 3 mm
* Teeth with mobility less than 0.5 mm
* Patients experiencing moderate (55-113 mm) or severe pain (114-170 mm) according to the Heft-Parker Visual Analog Scale (HP-VAS)

Exclusion Criteria:

* Patients with any systemic disease
* Teeth with open apex or radiographic evidence of periapical pathology
* Teeth showing internal or external root resorption
* Teeth that do not meet Glickman's periodontal health criteria or have probing depth > 3 mm
* Teeth with mobility greater than 0.5 mm
* Patients experiencing no pain (0 mm) or mild pain (1-54 mm) on the HP-VAS

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Success Rate of Mandibular Anesthesia | Within 30 minutes after anesthesia administration, during the endodontic procedure
  The success of inferior alveolar nerve block (IANB) will be determined based on the patient's pain response during endodontic treatment, measured using the Heft-Parker Visual Analog Scale (HP-VAS). Anesthesia will be considered successful if pain during treatment is rated as "none" or "mild" on HP-VAS.

SECONDARY OUTCOMES:
Correlation Between Dental Anxiety Level and Anesthesia Success | At the end of the single treatment session (within 30 minutes after anesthesia administration)
  Relationship between Modified Dental Anxiety Scale (MDAS; score range 5-25, higher scores indicate greater anxiety) and anesthesia success rates during a single endodontic treatment session.
Salivary Cortisol Level Change | Pre-anesthesia and 15 minutes post-anesthesia
  Difference in salivary cortisol levels measured 15 minutes before and 15 minutes after anesthesia to assess stress response related to dental anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Sciences University Faculty of Dentistry, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT07124273/Prot_SAP_000.pdf